CLINICAL TRIAL: NCT06225648
Title: The Threonine Requirement in Healthy Adults Over 60 Years
Brief Title: Threonine Requirement in Adults >60 Years of Age
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Glenda Courtney-Martin, Senior Associate Scientist, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1000081068
Record Dates: First submitted 2024-01-16; First posted 2024-01-26 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Healthy; Aging
Keywords: elderly; healthy; threonine requirement; indicator amino acid oxidation; stable isotopes
MeSH Terms: interventions — Threonine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Threonine in Adults > 60 (Experimental): Threonine: all subjects will receive up to 7 threonine test levels, in random order.
  Interventions: Other: threonine

INTERVENTIONS:
Other: threonine — There are 7 different threonine test levels ranging from 5 to 45 mg of threonine per kilogram body weight per day.

SUMMARY:
Threonine is an essential amino acid and must be obtained from the diet. The body's capacity to maintain adequate mucin synthesis is directly related to the bioavailability of certain amino acids, including threonine, serine and proline (1). Moreover, the rate of mucin synthesis has been demonstrated to be directly related to the availability of dietary threonine in healthy rats (2) and piglets (3,4). Intestinal inflammation is known to increase gastrointestinal threonine uptake and mucin synthesis in enterally fed minipigs (5). Additionally, in animals, mucin function/barrier has been shown to decline with age, leaving them more susceptible to bacterial penetration. Thus, with advancing age (6), a higher dietary supply of threonine may be needed for maintaining intestinal mucosal health. Despite this, the current threonine requirement is based on studies conducted exclusively in young adults. Thus, there is a need to determine the threonine requirement directly in older adults.

DETAILED DESCRIPTION:
To determine the threonine requirement in adults over the age of 60 years. With age, various physiological changes occur, including a decline in muscle and an increase in fat. Muscle reduction is a cause for concern as it may lead to weakness rendering regular daily activities more difficult.

The muscles in the human body are composed of proteins and those proteins are made of small building blocks termed amino acids. The human body has the ability to make some amino acids which are called the non-essential amino acids. However, there are specific amino acids that the body needs to make protein, but can only be supplied from the foods eaten. These are termed essential amino acids. Threonine is one of the essential amino acids. It is needed to synthesize mucins which are proteins that protect the gastrointestinal tract from bacterial invasion. The body's capacity to make mucins is directly related to the bioavailability of amino acids like threonine. However, evidence from animal data has shown that older mice have compromised mucus function compared to young mice leaving them more susceptible to bacterial penetration. Thus, a higher dietary supply of threonine may be needed for maintaining intestinal mucosal health as individuals age. The purpose of this study is to find out the threonine requirement in adults over 60 years using the minimally invasive Indicator Amino Acid Oxidation (IAAO) method.

ELIGIBILITY:
Inclusion Criteria:

* Consent provided
* Aged 60 to 90 years old
* In good general health as evidenced by medical history, physical health and blood draw
* Fasting blood glucose, hemoglobin A1c (HbA1c), urea, creatinine
* Willingness to participate in the study.
* BMI <30 kg/m2.

Exclusion Criteria:

* Presence of chronic disease and/or acute illness known to affect protein/amino acid metabolism (e.g. HIV, diabetes, cancer, liver or kidney disease, acute cold or flu)
* Taking medications known to affect protein/AA metabolism (e.g. steroids)
* Inability to tolerate the diet (i.e. allergy)
* Significant weight loss during the past month or consumption of weight reducing diets.
* Significant caffeine consumption (>2 cups per day)
* Significant consumption of alcohol (>1 drink per day i.e. 1 beer or ½ glass of wine).
* Unwilling to have blood drawn from a venous access, or using a ventilated hood indirect calorimeter for the purposes of the study.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-03 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Determination of threonine requirements in adults >60 years of age | up to 24 months
  To measure the threonine requirement investigators will collect breath samples from participants. From these samples, investigators will measure the amount of amino acids oxidized and how much is retained in the body when graded intakes of threonine are consumed by the participants consuming a controlled diet.

CONTACTS AND LOCATIONS:
Overall Officials: Glenda Courtney-Martin, MSc, PhD, RD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No